CLINICAL TRIAL: NCT02316873
Title: Rhythm and Music to Rehabilitate Reading Disorders
Acronym: ReMus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aix Marseille Université (Other)
Collaborators: WHO Collaborating Centre for Maternal and Child Health, Trieste (Other); University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Daniele Schon, PhD, Aix Marseille Université
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReMus R-11-85
Record Dates: First submitted 2014-12-09; First posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Reading Disability
Keywords: music training, rhythm
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music training (Experimental): twice a week one hour for 30 weeks, music training
  Interventions: Behavioral: Music training
- Visual arts (Active Comparator): twice a week one hour for 30 weeks, visual arts training
  Interventions: Behavioral: Visual arts

INTERVENTIONS:
Behavioral: Music training — This program was based on the Kodaly and Orff pedagogy and adapted to focus on rhythm and temporal processing.
  Arms: Music training
Behavioral: Visual arts — This program emphasized visual-spatial and hand skills as well as creativity.
  Arms: Visual arts

SUMMARY:
The purpose of this study is to determine whether music training is an effective treatment of reading disorders

DETAILED DESCRIPTION:
Introduction: Children with dyslexia show deficits in temporal processing, both in language and in music. Musical activity increases phonological awareness, word segmentation, working memory, as well as reading abilities in children with typical development, a compelling evidence for a role of music training in fostering brain plasticity. Within this theoretical framework, we investigate the hypothesis that music training, by improving temporal processing and rhythm abilities, improves phonological awareness and reading skills in children with dyslexia.

Methods: The study is a prospective, multicenter, open randomized controlled trial, consisting of test, rehabilitation and re-test

ELIGIBILITY:
Inclusion Criteria:

* Italian native language
* Reading performance (accuracy and/or speed) failed on at least two of three school grade standardized Italian tests: text, words, pseudowords (cut-offs: z-score <-1.8 standard deviations from the mean for speed scores, a score <5th percentile in the accuracy scores).
* Hearing and neurological examination within normal range
* Normal or corrected-to-normal visual acuity
* General IQ >85 at Wechsler Intelligence Scale for Children III.

Exclusion Criteria:

* Presence of comorbidity involving Attentional Deficit Disorders with Hyperactivity (ADHD)
* Presence of comorbidity involving Specific Language Impairment (SLI)
* Presence of comorbidity involving Oppositional Defiant Disorder (ODD)
* Severe emotional-relational impairments
* Previous formal musical or painting education for more than one year, other on-going treatment.
* Presence of other diseases (i.e. diabetes , cystic fibrosis, asthma...) that could influence the performance in cognitive and executive functions.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pseudoword reading test | six months
  The primary outcome variable was the performance in the pseudoword reading test measured in terms of accuracy (percentile of number of errors).

SECONDARY OUTCOMES:
Reading text | six months
  Reading a short standardized text, measured in terms of accuracy (percentile of number of errors) and speed (z score of reading syll/sec or time).
Phonological awareness | six months
  Phonemic blending task. Children have to blend sounds into words (e.g. hearing [c]-[a]-[t] and produce [cat]). The number of correct items is the dependent variable.
Word reading | six months
  The ability to read aloud single words and pseudowords is measured on a standardized list of 102 Italian words

REFERENCES:
- [Derived] Flaugnacco E, Lopez L, Terribili C, Montico M, Zoia S, Schon D. Music Training Increases Phonological Awareness and Reading Skills in Developmental Dyslexia: A Randomized Control Trial. PLoS One. 2015 Sep 25;10(9):e0138715. doi: 10.1371/journal.pone.0138715. eCollection 2015. PMID 26407242